CLINICAL TRIAL: NCT05247710
Title: Differential Mobility Spectrometry (DMS) Based Skin Tumor Analysis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tampere University Hospital (Other)
Collaborators: Olfactomics Oy (Unknown)
Responsible Party: Sponsor
Other Study IDs: R20100L
Record Dates: First submitted 2022-01-03; First posted 2022-02-21 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-04

CONDITIONS: Basal Cell Carcinoma
Keywords: Basal cell carcinoma (BCC); Differential mobility spectrometry (DMS); Automatic tissue analysis (ATAS)
MeSH Terms: conditions — Carcinoma, Basal Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Biospecimen Retention: Samples With DNA — * Punch biopsy (4 mm) of basal cell carcinoma tumor
  * Control biopsy (4 mm) of healthy skin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients diagnosed with non-superficial basal cell carcinoma
  Interventions: Procedure: Punch biopsy

INTERVENTIONS:
Procedure: Punch biopsy — Punch biopsy of basal cell carcinoma tumor and a control biopsy of healthy skin are collected during primary tumor excision surgery from each recruited patient.

SUMMARY:
The trial is a single-center, non-randomized feasibility study aiming to evaluate the feasibility of ex-vivo tissue analysis using differential mobility spectrometry (DMS) of tissue smoke generated by the use of an electrosurgical instrument.

Patients recruited in the trial receive standard-of-care basal cell carcinoma tumor excision surgery.

DETAILED DESCRIPTION:
Basal cell carcinoma (BCC) is the most common cancer in Caucasians and the average risk of developing BCC is approximately 30% (1,2). In Finland, BCC is the most common cancer and the incidence of BCC is approximately 49/100 000 in men and 45/100 000 in women (3).

There are several types of BCC (4) of which superficial type can be managed with non-operative treatment. All the other types of BCC (micronodular, nodular, infiltrative) require operative treatment which means surgical removal of the tumor with a few millimeters healthy skin margin (5). The aim of the operative treatment is to remove the tumor entirely so that the healthy skin margins are as sparing as possible and that the functional and cosmetic outcomes are as satisfactory as possible. Margin positiveness leads to one or more reoperations which increase the risk of surgical complications.

Differential mobility spectrometry (DMS) based application called automatic tissue analysis (ATAS) can be utilized to identify tumor cells from healthy tissue. Tissue identification is done by analyzing tissue smoke that is generated by the use of an electrosurgical instrument called diathermy (6,7).

The objective of the trial is to test whether it is possible to identify BCC from normal skin by using ATAS. A 4mm punch biopsy of BCC tumor and a control biopsy of healthy skin will be collected from 30 - 40 patients undergoing BCC tumor excision. The biopsies will be examined in the research laboratory with ATAS to test tissue recognition.

ELIGIBILITY:
Inclusion Criteria:

* Punch biopsy diagnosed basal cell carcinoma.
* Tumor diameter of 1,5 cm or larger.
* Operable patient that is willing to participate in the trial.

Exclusion Criteria:

* Tumor diameter of less than 1,5 cm.
* Patient that is unsuitable to take part in the trial, for example, has a tendency to develop keloids.
* Patient that is unwilling to take part in the trial.
* Patient that is not able to understand given information concerning the trial or to give consent to take part in the trial.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with non-superficial basal cell carcinoma and treated in the outpatient clinic of otorhinolaryngology in Tampere University Hospital, Finland.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-12-09 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Resolution of normal and cancerous tissue | Through study completion, an average of 1 year
  The ATAS device records a molecular spectrum of the surgical smoke generated when the collected tissue samples are processed with an electrosurgical instrument in the research laboratory. The primary outcome of the study is to test the ability of the device to correctly distinguish cancerous tissue from normal tissue based on predicted differences in the spectrum.

SECONDARY OUTCOMES:
Differentiation of basal cell carcinoma histopathological sub-types | Through study completion, an average of 1 year
  There are several histopathological sub-types of BCC which have a different kind of tumor growth. It is possible that the differences in tumor histopathology have an effect on the resolution of tissue types.
The influence of basal cell carcinoma tumor thickness and infiltration depth on the resolution | Through study completion, an average of 1 year
  BCC can grow nodularly forming a round-shape tumor, infiltratively through the layers of the skin causing ulcers and/or flatly. Each BCC tumor has one or more features in tumor growth. The overall thickness of the tumor and the infiltration depth of the tumor, both presented in millimetres, can have an effect on the resolution of tissue types.

CONTACTS AND LOCATIONS:
Overall Officials: Niku Oksala, M.D., Ph.D., Study Director — Tampere University Hospital
Locations (1):
- Tampere University Hospital, Tampere, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] English DR, Kricker A, Heenan PJ, Randell PL, Winter MG, Armstrong BK. Incidence of non-melanocytic skin cancer in Geraldton, Western Australia. Int J Cancer. 1997 Nov 27;73(5):629-33. doi: 10.1002/(sici)1097-0215(19971127)73:53.0.co;2-z. PMID 9398037
- [Background] Gallagher RP, Hill GB, Bajdik CD, Fincham S, Coldman AJ, McLean DI, Threlfall WJ. Sunlight exposure, pigmentary factors, and risk of nonmelanocytic skin cancer. I. Basal cell carcinoma. Arch Dermatol. 1995 Feb;131(2):157-63. PMID 7857111
- [Background] Hannuksela-Svahn A, Pukkala E, Karvonen J. Basal cell skin carcinoma and other nonmelanoma skin cancers in Finland from 1956 through 1995. Arch Dermatol. 1999 Jul;135(7):781-6. doi: 10.1001/archderm.135.7.781. PMID 10411152
- [Background] Sexton M, Jones DB, Maloney ME. Histologic pattern analysis of basal cell carcinoma. Study of a series of 1039 consecutive neoplasms. J Am Acad Dermatol. 1990 Dec;23(6 Pt 1):1118-26. doi: 10.1016/0190-9622(90)70344-h. PMID 2273112
- [Background] Bichakjian CK, Alam M. Reply to: "Comment on 'Guidelines of care for the management of basal cell carcinoma'". J Am Acad Dermatol. 2018 Nov;79(5):e101. doi: 10.1016/j.jaad.2018.06.051. Epub 2018 Jul 5. No abstract available. PMID 29981388
- [Background] Covington JA, van der Schee MP, Edge AS, Boyle B, Savage RS, Arasaradnam RP. The application of FAIMS gas analysis in medical diagnostics. Analyst. 2015 Oct 21;140(20):6775-81. doi: 10.1039/c5an00868a. PMID 26205889
- [Background] Sutinen M, Kontunen A, Karjalainen M, Kiiski J, Hannus J, Tolonen T, Roine A, Oksala N. Identification of breast tumors from diathermy smoke by differential ion mobility spectrometry. Eur J Surg Oncol. 2019 Feb;45(2):141-146. doi: 10.1016/j.ejso.2018.09.005. Epub 2018 Oct 15. PMID 30366874